CLINICAL TRIAL: NCT05284019
Title: An Exploratory, Prospective, Randomized, Pragmatic Open Label Cohort Study to Evaluate the Comparative Effectiveness of Eptinezumab in the United States
Brief Title: Real World Effectiveness of Eptinezumab in Participants With Migraine
Acronym: EVEC
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was terminated due to enrolment challenges.
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19766N
Record Dates: First submitted 2022-02-23; First posted 2022-03-17 (Actual); Results first posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — eptinezumab; erenumab; Botulinum Toxins, Type A; fremanezumab; galcanezumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Eptinezumab (Experimental): Participants will receive eptinezumab via intravenous (IV) infusion on Day 0 and Day 84.
  Interventions: Drug: Eptinezumab
- Anti-CGRP injectables (Experimental): Participants are free to select treatment from one of 3 calcitonin gene-related peptide (CGRP) inhibitors: erenumab, fremanezumab, or galcanezumab. CGRP inhibitors will be administered via subcutaneous (SC) injection on Day 0 and then, per product label.
  Interventions: Drug: Erenumab; Drug: Fremanezumab; Drug: Galcanezumab
- Onabotulinumtoxin-A (Experimental): Onabotulinumtoxin-A will be administered via intramuscular (IM) injection on Day 0 and Day 84.
  Interventions: Drug: Onabotulinumtoxin-A

INTERVENTIONS:
Drug: Eptinezumab — Concentrate for solution for IV infusion
  Other Names: Vyepti
  Arms: Eptinezumab
Drug: Erenumab — Solution for SC Injection
  Other Names: Aimovig®
  Arms: Anti-CGRP injectables
Drug: Onabotulinumtoxin-A — Solution for IM Injection
  Arms: Onabotulinumtoxin-A
Drug: Fremanezumab — Solution for SC Injection
  Other Names: Ajovy®
  Arms: Anti-CGRP injectables
Drug: Galcanezumab — Solution for SC Injection
  Other Names: Emgality®
  Arms: Anti-CGRP injectables

SUMMARY:
The purpose of this study is to examine how eptinezumab compares to other advanced preventive medications in a real-world community setting in adult participants with episodic migraine (EM) or chronic migraine (CM). These objectives include exploring the comparative effectiveness on patient reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of migraine per International Headache Society (IHS) International Classification of Headache Disorder (ICHD)-3 guidelines at least 12 months prior to screening.
* Have a history of ≥ 8 migraine days/month in 2 of the previous 3 months as confirmed by the treating physician through medical records.
* Be able to understand the clinical description of treatment options and have the capability to participate fully in making their treatment preferences known.
* Be willing to accept randomization to any of the possible study medications if allocated to that treatment arm.
* Be willing and capable of completing daily reports and other participant reported outcome measures using a smartphone-based application.

Exclusion Criteria:

* The participant has a history of severe drug allergy or hypersensitivity, or known hypersensitivity or intolerance to either eptinezumab, erenumab, fremanezumab, galcanezumab or their excipients.
* The participant has previous history of use of any of the study drugs (for example, eptinezumab, Botox, erenumab, fremanezumab or galcanezumab). Note that only previous Botox use for treatment of migraine is exclusionary. Prior use of Botox for cosmetic purposes is allowed.
* The participant has a diagnosis of CM and has hypersensitivity to botulinum toxin preparation or to any of the components in the formulation.
* The participant has used opioids or butalbital-containing products greater than 4 days per month in the last month.

Other inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-03-04 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2023-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (10):
- United States (10):
  - Gilbert Neurology Partners/ CCT Research, Gilbert, Arizona
  - Ki Clinical Research LLC, dba New England Institute for Clinical Research, Stamford, Connecticut
  - Innovation Medical Group, Palmetto Bay, Florida
  - The Headache Center, Ridgeland, Mississippi
  - StudyMetrix Research, City of Saint Peters, Missouri
  - North Kansas City Hospital, North Kansas City, Missouri
  - Dent Neurologic Institute - Amherst, Amherst, New York
  - Carolina Women's Research and Wellness Center, Durham, North Carolina
  - AIM Trials, LLC, Plano, Texas
  - Olympus Family Medicine/CCT Research, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Groups:
- Erenumab: Participants received erenumab SC every 28 days, as per the product label for 6 months.
- Fremanezumab: Participants received fremanezumab SC every 28 days or every 84 days, as per the product label for 6 months.
- Onabotulinumtoxin-A: Participants received onabotulinumtoxin-A SC at Baseline (Day 0) and Week 12.
- Galcanezumab: Participants received galcanezumab loading dose SC as applicable followed by dosing every 28 days, as per the product label for 5 months.
- Eptinezumab: Participants received eptinezumab via IV infusion, as per the product label at Baseline (Day 0) and Week 12.
Period: Overall Study
Arm/Group | Erenumab | Fremanezumab | Onabotulinumtoxin-A | Galcanezumab | Eptinezumab
Started | 3 | 2 | 2 | 8 | 17
Received at Least 1 Dose of Study Drug | 3 | 2 | 2 | 8 | 16
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 2 | 2 | 8 | 17
Not completed — Study terminated | 2 | 2 | 2 | 5 | 15
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Erenumab | Fremanezumab | Onabotulinumtoxin-A | Galcanezumab | Eptinezumab | Total
Number analyzed (Participants) | 3 | 2 | 2 | 8 | 17 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.3 (6.4) | 60.5 (4.9) | 30.5 (17.7) | 43.1 (12.6) | 38.2 (10.5) | 41.2 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 2 | 6 | 15 | 28
  Male | 0 | 0 | 0 | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 0 | 1 | 5 | 9
  Not Hispanic or Latino | 1 | 1 | 2 | 7 | 12 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 4 | 4 | 10
  White | 3 | 1 | 1 | 4 | 12 | 21
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Patient-informed Most Bothersome Symptom (PI-MBS) Score at Week 24
Description: Participants select the symptom that they find most impairs them at the time of reporting and rate the severity of that symptom on a 7-point scale (1 = very much improved; 2 = much improved; 3 = minimally improved; 4 = no change; 5 = minimally worse; 6 = much worse; 7 = very much worse) where a high score indicated worsening. Score ranges from 1 (Very Much Improved) to 7 (Very Much Worse). Lower scores indicate better health status. The MBS areas included: nausea, vomiting, sensitivity to light, sensitivity to sound, mental cloudiness, fatigue, pain with activity, mood changes, and other symptoms.
Time Frame: Baseline, Week 24
Population: Analysis was performed on the full analysis set (FAS), which included all participants who completed at least one daily report after receiving eptinezumab or other advanced migraine therapy. Due to the small sample size, data was not reported for participant confidentiality reasons.
Arm/Group | Erenumab | Fremanezumab | Onabotulinumtoxin-A | Galcanezumab | Eptinezumab
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of "Good Days" From Baseline
Description: The participants report the number of "good days" and "bad days" they had in the previous week on a weekly basis using the good day/bad day scale.
Time Frame: Up to Week 24
Population: Analysis was performed on the FAS, which included all participants who completed at least one daily report after receiving eptinezumab or other advanced migraine therapy. Due to the small sample size, data was not reported for participant confidentiality reasons.
Arm/Group | Erenumab | Fremanezumab | Onabotulinumtoxin-A | Galcanezumab | Eptinezumab
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Change From Baseline in Quality of Life (QOL) as Measured by the 5 Level Euro Quality of Life 5 Dimensional Questionnaire (EQ-5D-5L) Score at Week 24
Description: The EQ-5D-5L is a participant-reported assessment designed to measure the participant's well-being. It consists of 5 descriptive items (mobility, self-care, usual activities, pain/discomfort, and depression/anxiety) and a visual analog scale (VAS) of the overall health state. Each descriptive item is rated on a 5-point index ranging from 1 (no problems) to 5 (extreme problems). The VAS ranges from 0 (worst imaginable health state) to 100 (best imaginable health state).
Time Frame: Baseline, Week 24
Population: as for outcome 2
Arm/Group | Erenumab | Fremanezumab | Onabotulinumtoxin-A | Galcanezumab | Eptinezumab
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Health Care Resources Utilization (HCRU): Number of Participants Who Used Health Services and Medications
Time Frame: Up to Week 24
Population: as for outcome 2
Arm/Group | Erenumab | Fremanezumab | Onabotulinumtoxin-A | Galcanezumab | Eptinezumab
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: QOL as Measured by the 6 Item Headache Impact Test (HIT-6) Score
Description: The HIT-6 (version 1.0) is a Likert-type, self-reporting questionnaire designed to assess the impact of an occurring headache and its effect on the ability to function normally in daily life. The HIT-6 contains 6 questions, each item is rated from never to always with the following response scores: never = 6, rarely = 8, sometimes = 10, very often = 11, and always = 13. The total score for the HIT-6 is the sum of each response score ranging from 36 to 78. The life impact derived from the total score is described as follows: severe (≥60), substantial (56-59), some (50-55), little to none (≤49).
Time Frame: Up to Week 24
Population: as for outcome 2
Arm/Group | Erenumab | Fremanezumab | Onabotulinumtoxin-A | Galcanezumab | Eptinezumab
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: QOL as Measured by the Migraine Disability Assessment (MIDAS) Total Score
Description: The Midas score is a participant completed 5-item questionnaire about lost time and productivity (for work, school or family/social activities) in the past 3 months (number of days missed) where: 0-5=Little or No disability, 6-10=Mild disability, 11-20=Moderate disability or 21+ Severe disability.
Time Frame: Up to Week 24
Population: as for outcome 2
Arm/Group | Erenumab | Fremanezumab | Onabotulinumtoxin-A | Galcanezumab | Eptinezumab
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Participant Satisfaction Score as Measured by the Treatment Satisfaction Questionnaire for Medication (TSQM)
Description: The TSQM assesses four domains of participants' satisfaction with treatment, with scale ranges from 0 (extremely dissatisfied) to 100 (not at all dissatisfied) for each of the categories (Effectiveness, Side Effects, Convenience, and Overall Satisfaction).
Time Frame: Week 24
Population: as for outcome 2
Arm/Group | Erenumab | Fremanezumab | Onabotulinumtoxin-A | Galcanezumab | Eptinezumab
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Percentage of Participants That Switch From the Preventive Medication They Are Randomized to at Baseline to Another Preventive Medication
Time Frame: Week 24
Population: as for outcome 2
Arm/Group | Eptinezumab | Onabotulinumtoxin-A | Erenumab | Fremanezumab | Galcanezumab
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Week 24
Description: The safety population included all participants who received treatment.
Arm/Group | Erenumab | Fremanezumab | Onabotulinumtoxin-A | Galcanezumab | Eptinezumab
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2 | 0/2 | 0/8 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2 | 0/2 | 0/8 | 0/16
Other Adverse Events (participants affected / at risk) | 0/3 | 0/2 | 0/2 | 6/8 | 4/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erenumab (N=3) | Fremanezumab (N=2) | Onabotulinumtoxin-A (N=2) | Galcanezumab (N=8) | Eptinezumab (N=16)
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Pelvic floor dysfunction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 1
Swelling face (General disorders) | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Attention deficit hyperactivity disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The study was terminated early due to enrolment challenges.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-07-07): https://cdn.clinicaltrials.gov/large-docs/19/NCT05284019/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-04): https://cdn.clinicaltrials.gov/large-docs/19/NCT05284019/SAP_001.pdf